CLINICAL TRIAL: NCT06617286
Title: MAC-CAR: a Phase 1B/II Trial of Myeloablative Conditioning and Autologous Stem Cell Transplantation Followed by Autologous CD30+ CAR T Cells in Children, Adolescents and Young Adults with Poor-Risk Classical Hodgkin Lymphoma (cHL)
Brief Title: CD30 CAR T-cells Post AutoHSCT for Poor-risk Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 624
Record Dates: First submitted 2024-09-09; First posted 2024-09-27 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: classical Hodgkin lymphoma; CAR T-cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD30 CAR T-cells (Experimental): Patients will receive autologous CD30 CAR T-cells post autologous stem cell transplant between days 21-42.
  Interventions: Biological: CD30 CAR T-cell

INTERVENTIONS:
Biological: CD30 CAR T-cell — After MAC and AutoHSCT patients will receive CD30+ CAR T-cells (Phase 1B dose level 1 - 1x108/m2 (max 2.5x108) or dose level 2 - 2x108/m2 (max 5.0 x108) 21-42 days after the AutoHSCT and the RP2D dose level obtained in the Phase IB part administered in the Phase II portion.

SUMMARY:
Patients with poor risk classical Hodgkin Lymphoma (cHL) will undergo myeloablative chemotherapy (MAC) with autologous stem cell transplantation (AutoHSCT) and subsequently receive autologous CD30+ CAR T-cells.

DETAILED DESCRIPTION:
Eligible patients will be screened for study entry and proceed to cell procurement at local sites with collection of peripheral blood mononuclear cells (PBMC) for CD30+ CAR T-cell manufacturing at UNC. Patients will then have autologous stem cells collected (PBSC) and stored for future AutoHSCT.

After another screening for MAC+AutoHSCT, patients who meet criteria will receive BEAM conditioning followed by AutoHSCT. About 21-42 day after the autologous stem cell infusion, patients will receive their autologous CD30+ CAR T-cell infusion, if they meet subsequent pre CD30+ CAR T-cell eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥ 6 and ≤ 29.99 years at the time of consent.
* Lansky OR Karnofsky score of ≥ 60% (see Appendix VI)
* Disease Status: Confirmed diagnosis of CD30+ classical Hodgkin Lymphoma and meets eligibility to undergo ASCT. Must meet one of the following:

Induction failure Progressive disease Disease relapse (1st, 2nd or 3rd)

* Confirmatory re-biopsy of relapse/refractory/persistent CD30+ cHL prior to study entry.
* Risk Factors: Patient must meet 2 or more of the established risk factors:

Performance score (Karnofsky/Lansky) <;90% Time from diagnosis to first relapse of <1 year Extra nodal involvement at the time of relapse/progression High baseline metabolic tumor volume (MTV, >60mL) by 18F-fluorodeoxyglucose positron emission tomography (PET)/computed tomography (CT) Chemo resistant disease (Deauville 4-5) after the first re-induction

Exclusion Criteria:

* not meeting the inclusion criteria

Ages: 6 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2039-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of administering CAR T-cells | 2 years
  To evaluate the incidence of adverse events related to autologous CD30+ CAR T-cell infusions including not limited to infusions related reactions (IRR) (CTCAE 5.0), cytokine release syndrome (CRS) (ASCTC), and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) (ASCTC) and all general grade 3-5 toxicities (CTCAE 5.0) in children, adolescent, and young adult patients with poor-risk CD30+ cHL following MAC AutoHSCT.
Feasibility of Central Manufacturing of CAR T-cells | 1 year
  To evaluate the feasibility of local site PBMC collection and central GMP CD30 CAR T cell manufacturing with a 75% success rate in children, adolescent, and young adult patients with poor-risk CD30+ cHL following MAC AutoHSCT.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided